CLINICAL TRIAL: NCT03025464
Title: Wireless Sensor Patch for Educing Barriers to In-home Sleep Apnea Screening, Phase II
Brief Title: Validation of Sleep Apnea Screening Device Phase II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued prematurely due to funding insecurity
Sponsor: University of Michigan (Other)
Collaborators: Zansors (Industry)
Responsible Party: Principal Investigator, J. Todd Arnedt, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R42MD008845-02 (NIH)
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Obstructive Sleep Apnea Screening Device — Assessment of ability of device to detect apneas and hypopneas to screen for OSA

SUMMARY:
Obstructive sleep apnea (OSA) is the most common type of sleep apnea. The marketplace currently does not have an affordable, easy-to-use, over-the-counter, home-based OSA screening device. An affordable, available, FDA-approved and easy-to-use over-the-counter OSA screening tool would allow greater screening of at-risk individuals, especially in underserved communities with low socioeconomic status, hopefully encouraging a greater proportion of such individuals to seek treatment for their condition. Over the past year, this investigative team has engineered a small screening device (Zerify®) for OSA and obtained preliminary evidence of its efficacy in a clinical population under a NIMHD-sponsored Phase I STTR award. Phase I Specific Aims 1 and 2 focused on developing a small (1.5 x 2.5 x 0.2 inches) semiconductor sensor that could store sound/motion data, transfer these data to a computer, and detect non-clinical simulated apnea events with a specificity and specificity exceeding 90%. Phase I Specific Aim 3 established the preliminary psychometric performance data of the screening device in a clinical sample of 52 patients (13% African American, 6% Asian, 4% Mixed or Other Race) against gold-standard polysomnography. Phase II proposal aims to optimize the engineered hardware and associated OSA algorithms, create a patient companion app and wireless healthcare provider dashboard, and compare the efficacy of this screening device to the most commonly utilized sleep apnea screener, the home sleep apnea test (HSAT).

DETAILED DESCRIPTION:
An alternative to polysomnography (PSG), which is done overnight in a lab, is home sleep apnea testing (HSAT). Also known as out-of-center testing, HSAT has emerged as a more convenient and increasingly widely used method to screen for sleep apnea. HSAT records fewer signals for assessment, is less cumbersome than traditional PSG, and allows patients to spend the night at home, eliminating the need for technical staff to be present during testing. HSAT is considerably less expensive than PSG to perform. Despite its advantages, there are concerns about false-negatives and underestimation of disease severity with HSAT. There is clearly a need to improve the accuracy of less costly screening tools for OSA. Zansors® wireless microsensor is a novel device to screen for sleep apnea, which measures breathing patterns and movement, and which will collect data and communicate with a smartphone via Bluetooth. In this study, investigators are comparing the Zansors microsensor to HSAT and PSG to assess its accuracy. Patients will be asked to wear the device during the clinical HSAT ordered by their doctor, and again at an in-laboratory sleep study. When patients are being trained to use the HSAT equipment, research staff will also show them how to put the Zansors® device on. They will then wear it at home on the night of their HSAT. At a later date, when they come for the in-laboratory sleep study, the device will again be worn overnight while they are being assessed by the full PSG equipment. Together in this study, all these device recordings will help to detect any sleep apnea and researchers will compare the results of the Zansors ® microsensor with HSAT and PSG equipment. If the Zansors ® device is confirmed to detect sleep hypopneas and apneas accurately, it can be used easily and inexpensively by people at home to screen for obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 and referred by medical staff for an assessment for suspected sleep apnea using either a home sleep apnea testing device or in-lab PSG equipment

Exclusion Criteria:

* Pregnancy
* Heart disease including congestive heart failure or a pacemaker
* Breathing disorder (emphysema or chronic obstructive breathing disorder)
* Neurological disorder such as Parkinson's Disease
* Restless leg syndrome or Periodic limb movement
* Allergies to metal
* Pre-existing skin conditions where sensor would be attached

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Specificity | 8 hours
  Specificity of Zansors' device to detect hypopneas and apneas compared to home sleep apnea test devices and to polysomnography over an 8-hour period of sleep at 30-second intervals.

SECONDARY OUTCOMES:
Sensitivity | 8 hours
  Sensitivity of Zansors' device to detect hypopneas and apneas compared to home sleep apnea test devices and to polysomnography over an 8-hour period of sleep at 30-second intervals.
Positive Predictive Value (PPV) | 8 hours
  PPV of Zansors' device to detect hypopneas and apneas compared to home sleep apnea test devices and to polysomnography over an 8-hour period of sleep at 30-second intervals.
Negative Predictive Value (NPV) | 8 hours
  NPV of Zansors' device to detect hypopneas and apneas compared to home sleep apnea test devices and to polysomnography over an 8-hour period of sleep at 30-second intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No